CLINICAL TRIAL: NCT03506919
Title: Comparative Clinical Efficacy and Safety of Coded Polyherbal Medicine Arthitec 1 and Arthitec 2 With Allopathic Medicine for the Management of Arthritis
Brief Title: Comparative Clinical Efficacy and Safety of Coded Polyherbal Medicine for the Management of Arthritis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shifa Ul Mulk Memorial Hospital (Other)
Responsible Party: Principal Investigator, Hafiz Muhammad Asif, Assistant Professor, Shifa Ul Mulk Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 003
Record Dates: First submitted 2018-01-12; First posted 2018-04-24 (Actual); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Treatment of Arthritis
MeSH Terms: interventions — Allopurinol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arthitec 1 (Experimental)
  Interventions: Drug: Allopurinol
- Arthitec 2 (Experimental)
  Interventions: Drug: Allopurinol

INTERVENTIONS:
Drug: Allopurinol — Allopurinol is used to treat gout and certain types of kidney stones. It is also used to prevent increased uric acid levels in patients receiving cancer chemotherapy. These patients can have increased uric acid levels due to release of uric acid from the dying cancer cells. Allopurinol works by reducing the amount of uric acid made by the body. Increased uric acid levels can cause gout and kidney problems

SUMMARY:
This study aimed to develop two poly herbal capsule formulations for arthritis through granulation and conduction of their clinical trial in order to achieve quality, efficacy and safety. Arthritis is a chronic disease of unknown cause. An inflammatory disease of the synovium, it results in pain, stiffness, swelling, deformity and, eventually, loss of function in the joints. Despite early detection, current treatment medications are limited in their efficacy and are frequently toxic. Many patients look for complementary and alternative medicine (CAM) options in coping with this debilitating disease. Research has indicated that people suffering from chronic pain, as in arthritis, and those dissatisfied with current treatment are very likely to seek alternative treatments, and an estimated 60-90% of persons with arthritis use complementary and alternative medicines. Among the most widely used treatments are chiropractic and herbal therapies. This growing interest in alternative medical practices clearly indicates the need for more thorough investigation into the safety and efficacy of herbal medicine. Thousand years of traditional use can provide us with valuable guidelines to the selection, preparation and application of herbal formulation. To be accepted as viable alternative to modern medicine, the same vigorous method of scientific and clinical validation must be applied to prove the safety and effectiveness of a therapeutical product.

DETAILED DESCRIPTION:
Although there are more than 100 different kinds of arthritis, the three most common are gout, osteoarthritis (OA) and rheumatoid arthritis (RA).Gout occurs in response to the presence of monosodium urate (MSU) crystals in joints, bones and soft tissues, and is usually treated by non-steroidal anti-inflammatory drugs (NSAIDs), oral or intravenous colchicines, and oral, intravenous or intraarticular glucocorticoids. All these drugs can abort acute attacks, but they also may have severe side effects. OA results from articular cartilage failure induced by a combination of genetic, metabolic, biochemical and biomechanical factors. OA is normally treated with analgesics such as acetaminophen and opioids, NSAIDs, and intraarticular therapies such as glucocorticoids and hyaluronans.

In RA, 75% of the sufferers are women, suggesting the importance of hormones in the etiology of the disease. Smoking and stress are also thought to contribute to this disease, which is characterized by joint stiffness and swelling, often in a symmetrical pattern on both sides of the body. The goals of management of patients with RA are to control pain and swelling, delay disease progression, minimize disability, and improve quality of life. For pain control and swelling, treatment includes analgesics such as acetaminophen and opioids, NSAIDs, and intra-articular therapies such as glucocorticoids. In addition, disease modifying anti-rheumatic drugs (DMARDs) are used to modify the clinical and radiological course of RA. Examples include methotrexate (MTX), sulfasalazine, leflunomide, hydroxychloroquine and newer therapies such as anti-tumor necrosis factor (TNF)-a therapy (etanercept, infliximab and adalimumab), anti-CD20 therapy (rituximab) and abatacept However, all of these agents are associated with numerous side effects Promising evidence has been found for the effective use of some herbal preparations in the treatment of arthritis. Furthermore, evidence suggesting that some herbal preparations reduce consumption of non-steroidal anti-inflammatory drugs. It has been evident that some herbal preparations (Tripterygium wilfordii Hook F) monotherapy is not inferior then methotrexate and in combination with methotrexate showed better result than alone. In addition, adverse effect associated with trials of herbal preparation for arthritis is not only fewer but also minor. Evidence-based complementary and alternative medicine treatments are remarkably successful in addressing not only chronic but acute health issues as well. It is strongly perceived that different complementary and alternative medicine treatments exerts their healing potential by influencing immune system.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from Arthritis

Exclusion Criteria:

* Patients with Hypertension, Cardiovascular disorders and Kidney disorders were excluded

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-04-30 (Estimated); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
Reduction in Serum Uric Acid level | 8 weeks
  Reduction in Serum Uric Acid level will be monitored after 8 weeks. Increase level of Serum Uric acid is the major cause of Gouty arthritis which is more prevalent in South-Asian countries.

CONTACTS AND LOCATIONS:
Locations (1):
- clinical trial was conducted in Bahawalpur, and Rawalpindi, Bahawalpur, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided